CLINICAL TRIAL: NCT00055016
Title: Registry of Fabry Disease: A Multicenter, Longitudinal Observational Study
Brief Title: Registry of Fabry Disease - A Multicenter Observational Study
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke@@@Shire Human Genetic Therapies (HGT) (Unknown)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030106; 03-N-0106
Record Dates: First submitted 2003-02-15; First posted 2003-02-17 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-03-03

CONDITIONS: Fabry Disease
Keywords: Lysosomal Disease; Renal Function; Stroke; Cardiac Disease; Natural History; Fabry Disease
MeSH Terms: conditions — Fabry Disease; Stroke; Heart Diseases

SUMMARY:
The purpose of this study is to compile a registry of patients with Fabry disease, an inherited metabolic disorder. In this disease, an enzyme called a-galactosidase A, which normally breaks down a lipid (fatty substance) called globotriaosylceramide (Gb3), is missing or does not function properly. As a result, Gb3 accumulates, causing problems with the kidneys, heart, nerves, and blood vessels. It is not known exactly how lipid accumulation causes these problems, but in another lipid storage disease called Gaucher disease the illness can be reversed if the accumulated lipid is removed by repeated intravenous (into a vein) infusions of the deficient enzyme.

The Fabry disease registry is a voluntary and anonymous list of patients that includes information about their health and allows doctors to follow changes in their symptoms and test results over time. It also allows doctors to compare symptoms between patients who are receiving certain therapies with those who are not receiving therapy. The goals of the registry are to:

* Better understand the natural history of Fabry disease, including disease variations within and between affected families;
* Provide a basis for developing guidelines for disease management;
* Evaluate how treatment affects the course of disease;
* Provide high-quality data and analyses that will help to continuously develop better treatments.

Patients of all ages with biochemical or genetic evidence of Fabry disease (i.e., individuals who have a deficiency of the enzyme a-galactosidase A or a mutation in the gene that encodes this enzyme, or both) are eligible for this study. This worldwide study will include 100 patients participating in Fabry disease studies at the NIH. These patients will come to the NIH Clinical Center only as required for participation their Fabry disease study. No additional procedures will be required for the current registry study.

NIH patients will take part in the registry study for their lifetime, or as long as they are being followed at the NIH for their Fabry disease. At their regularly scheduled NIH clinic visits, participants will have routine medical procedures and examinations deemed necessary by the doctor. The results of blood and urine tests taken at these visits will be entered into the registry database. Blood tests will include information on genotype (determination of which gene mutation is responsible for the disease), a-galactosidase A levels, Gb3 levels, and creatinine. Urine tests results will include creatinine clearance (a measure of kidney function) and protein evaluation.

DETAILED DESCRIPTION:
PROTOCOL TITLE: Registry of Fabry Disease: A Multicenter, Longitudinal Observational Study

PROTOCOL IDENTIFIER: FOS (Fabry Outcome Survey)

PHASE OF DEVELOPMENT: Post Marketing Outcome Survey (Outcome Survey)

SURVEY OBJECTIVES/ENDPOINTS:

The primary objectives of this outcome survey are to:

* enhance the understanding of the natural history of Fabry disease, including the intra- and inter-familial variations
* provide a basis for the development of management guidelines for Fabry disease
* evaluate the impact of therapeutic intervention on the clinical course of Fabry disease
* generate data and analyses to enable the continuous improvement of Fabry disease treatment
* collect long term safety and efficacy data on patients treated with Replagal enzyme replacement therapy

INCLUSION CRITERIA:

This registry/outcome survey is open for all patients of all ages, male and female, with a confirmed diagnosis of Fabry disease.

EXCLUSION CRITERIA:

* Patients who are unwilling to give informed consent.
* Patients who are receiving enzyme replacement therapy other than Replagal for Fabry Disease
* Patients currently enrolled in an ongoing blinded clinical trial in which the product is considered investigational.

NUMBER OF SUBJECTS PLANNED AND DURATION OF SUBJECT PARTICIPATION:

There is no predetermined number of patients that must be enrolled into the outcome survey. Patients who have been diagnosed (biochemically or genetically) with Fabry disease that consent to participate will be followed for an undetermined amount of time (i.e., until the sponsor closes the outcome survey or the patient withdraws consent).

TREATMENTS ADMINISTERED AND TREATMENT SCHEDULE:

Patients consenting to participate in the outcome survey will either be untreated or treated with Replagal ERT. It is recommended that patients be followed at increments determined to be necessary by the treating physician. It is also recommended that data on all patients be entered into the outcome survey on a bi-annual basis (every six (6) months).

Patients will not be supplied with Replagal at no charge as a result of participating in the Fabry Outcome Survey (FOS). Patients will receive Replagal through their participation in ongoing open label clinical trials or compassionate programs. Additionally, patients may receive commercially available product.

SURVEY ASSESSMENT SCHEDULE:

It is recommended that patients be followed at clinically relevant intervals determined by their treating physician. Data collected is to be entered into the FOS database as soon as possible after physician assessments.

SURVEY METHODOLOGY:

Observational data will be recorded in the FOS database based on routine clinical evaluations performed by the treating physician.

STATISTICAL METHODOLOGY:

The statistical analysis of FOS data will be performed by a bio-statistician designated by Shire HGT and in accordance with documented company guidelines and standard operating procedures.

ELIGIBILITY:
* INCLUSION CRITERIA:

This registry is open for all patients of all ages, male and female, with a confirmed diagnosis of Fabry disease.

EXCLUSION CRITERIA:

Patients who are unwilling to give informed consent.

Patients who are receiving enzyme replacement therapy other than Replagal for Fabry Disease.

Patients currently enrolled in an ongoing blinded clinical trial in which the product is considered investigational.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2003-02-13; Study Completion 2008-03-03

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Transkaryotic Therapies, Inc., Cambridge, Massachusetts

REFERENCES:
- [Background] Kaye EM, Kolodny EH, Logigian EL, Ullman MD. Nervous system involvement in Fabry's disease: clinicopathological and biochemical correlation. Ann Neurol. 1988 May;23(5):505-9. doi: 10.1002/ana.410230513. PMID 3133979